CLINICAL TRIAL: NCT02835430
Title: Coronally Advanced Flap and PRF With or Without Demineralized Freeze-dried Bone Allograft in Gingival Recession
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dr. D. Y. Patil Dental College & Hospital (Other)
Responsible Party: Principal Investigator, POONAM DHOLAKIA, Dr. Poonam Dholakia, Dr. D. Y. Patil Dental College & Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DPU/831(11)/2014
Record Dates: First submitted 2016-07-09; First posted 2016-07-18 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Gingival Recession
Keywords: Coronally advanced flap; Gingival recession; Bone, demineralized; Bone, freeze-dried; platelet-rich fibrin; root coverage procedures
MeSH Terms: conditions — Gingival Recession; Bone Diseases, Metabolic | interventions — Prolactin-Releasing Hormone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Coronally advanced flap and PRF with DFDBA (Experimental): Coronally advanced flap and platelet-rich fibrin membrane with demineralized freeze-dried bone allograft.
  Interventions: Procedure: Coronally advanced flap and PRF with DFDBA
- Coronally advanced flap and PRF without DFDBA (Active Comparator): Coronally advanced flap and Platelet-rich fibrin membrane without demineralized freeze-dried bone allograft.
  Interventions: Procedure: Coronally advanced flap and PRF without DFDBA

INTERVENTIONS:
Procedure: Coronally advanced flap and PRF with DFDBA — • For Test site: i. Following pre-suturing of coronally advanced flap, DFDBA (Rocky Mountain Particulate Allograft) was placed over the exposed root and adjacent bone surface and subsequently covered by PRF membrane.
  Other Names: Coronally advanced flap and Platelet-Rich Fibrin (PRF) with demineralized freeze-dried bone allograft (DFDBA Rocky Mountain Allograft)
  Arms: Coronally advanced flap and PRF with DFDBA
Procedure: Coronally advanced flap and PRF without DFDBA — . For Control site: i. Following pre-suturing of coronally avanced flap, exposed root and adjacent bone surface was covered by PRF membrane.
  Other Names: Coronally advanced flap and Platelet-Rich Fibrin (PRF) without demineralized freeze-dried bone allograft (DFDBA Rocky Mountain Allograft)
  Arms: Coronally advanced flap and PRF without DFDBA

SUMMARY:
* Gingival recession is defined as the apical migration of gingival margin beyond cemento-enamel junction with the exposure of root surface. More than 20% of the population presents one or more tooth surfaces with gingival recession.
* The main conditions leading to the development of this defect are gingival anatomical factors, chronic trauma, periodontitis, malposed tooth and dentinal hypersensitivity.
* The main goal of treating gingival recession is to restore the gingival margin to cement-enamel junction (CEJ) and normal sulcus with a functional attachment.
* A recent innovation in Guided Tissue Regeneration (GTR) technique is the use of second generation platelet concentrate, called as Platelet-Rich Fibrin membrane (PRF) that contains growth factors and cicatricial properties for root coverage procedures.
* Space is necessary to provide a channel for the migration of progenitor cells towards and on the denuded root surface, where they can differentiate into cementum and periodontal ligament cells.
* Since the gingival recession defects are non-space making, it may be difficult using the membrane technique alone, and hence, the use of a graft material underneath the membrane may help to resolve this problem. Root coverage tended to be better with the addition of demineralized freeze-dried bone allograft (DFDBA). These allografts prevent the collapse of membrane into the defect, stimulate the proliferation of osteogenic progenitor cells, and are thus, capable of promoting regeneration of attachment apparatus.
* Till date, no study is available in the literature on clinical evaluation of CAF (Coronally Advanced Flap)+PRF+DFDBA vs CAF+PRF for the management of gingival recession defects.
* And hence, this study is designed to evaluate the clinical efficacy of DFDBA (Rocky Mountain Particulate Allograft) for the management of isolated gingival recession defects.

DETAILED DESCRIPTION:
SURGICAL PROCEDURE:

I. After patient selection and obtaining informed consent, a total of 10 bilateral facial, Miller's Class I or II gingival recession defects were consecutively treated. Test and Control site were randomly assigned by flip coin technique.

II. The Test sites were treated using CAF+PRF+DFDBA and the Control sites were treated using CAF+PRF.

III. Under local anesthesia, an intrasulcular incision was given using a surgical bade on the buccal aspect of the involved tooth. The incision was extended horizontally to dissect the buccal aspect of the adjacent papillae, both mesially and distally, leaving the gingival margin of the adjacent teeth untouched. Two oblique releasing incisions were made from the mesial and distal extremities of the horizontal incision beyond the mucogingival junction.

IV. Partial-full-partial thickness flap was raised and extended beyond the mucogingival junction. The exposed root surface was thoroughly debrided and prepared to reduce the root convexities, if any.

V. A mesio-distal and apical dissection parallel to the vestibular lining mucosa was performed to release the residual muscle tension and facilitate the passive coronal displacement of the flap. The papillae adjacent to the involved tooth was de-epithelialized.

Preparation of PRF:

Preoperatively, a 10 ml of blood sample of the patient without anticoagulant was collected in a test tube and centrifuged immediately at 3000 rpm for 10 minutes. The platelet-rich fibrin clot was separated from the other two layers (acellular plasma and red blood cells) and prepared in the form of a membrane by squeezing out fluids from the fibrin clot.

. For Test site: i. Following pre-suturing, DFDBA (Rocky Mountain Particulate Allograft) was placed over the exposed root and adjacent bone surface and subsequently covered by PRF membrane.

ii. Flap was coronally displaced without tension and sutured using 4-0 mersilk non-resorbable suture.

iii. Additional lateral sutures were placed to close the releasing incisions.

. For Control site: i. Following pre-suturing, exposed root and adjacent bone surfaces were covered by PRF membrane.

ii. Flap was coronally displaced without tension and sutured using 4-0 mersilk non-resorbable suture.

iii. Additional lateral sutures were placed to close the releasing incisions.

Post-surgical protocols:

Postoperative instructions were given along with a recommendation to refrain from mechanical cleaning on the surgical areas. Periodontal dressing was placed at both Test and Control sites. Patients were instructed to apply 0.12% chlorhexidine solution (1:1 dilution) with a cotton swab twice daily for 14 days. Analgesics and antibiotics were prescribed and suture removal was performed 14 days post-surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age group of 18-45 years from both sexes.
* Presence of bilateral isolated gingival recession classified as Miller's class I or class II recession defects in anteriors and/or premolars.
* Systemically healthy patients.
* Patients willing to comply with all study-related procedures and available for follow-up.
* Ability to maintain good oral hygiene.

Exclusion Criteria:

* History of prolonged use of antibiotics/steroids/immunosuppressive agents/aspirin/ anticoagulants/other medications.
* Pregnant/Lactating women.
* Tobacco in any form.
* History of systemic diseases like hypertension, diabetes, HIV, bone metabolic disorders, radiation therapy, immunosuppressive therapy, cancer.
* Patients with unacceptable oral hygiene.
* Faulty tooth brushing technique.
* Malaligned teeth.
* Cervical abrasion.
* Unwilling patients.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2014-11; Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Recession Depth (RD) | Change from Baseline Recession Depth at 6 months.
  Recession depth (RD), measured from the cemento-enamel junction (CEJ) to the most apical extension of gingival margin at Baseline and 6 months post-surgery.

SECONDARY OUTCOMES:
Relative Attachment Level (RAL) | Change from Baseline Relative Attachment Level at 6 months.
  Relative Attachment Level from the lower border of stent to the base of sulcus at Baseline and 6 months post-surgery.
Probing Depth | Change from Baseline Probing Depth at 6 months.
  Probing depth was recorded from the crest of gingival margin to the base of gingival sulcus at Baseline and 6 months post-surgery.
Width of Keratinized Gingiva (WKG) | Change from Baseline Width of Keratinized Gingiva at 6 months.
  Width of Keratinized Gingiva (WKG) measured from the gingival margin to the mucogingival junction at Baseline and 6 months post-surgery.
Percentage of Root Coverage | At 6 months.
  (Preoperative recession depth - Postoperative recession depth)/ Preoperative recession depth * 100, at 6 months post-surgery.

REFERENCES:
- [Background] Padma R, Shilpa A, Kumar PA, Nagasri M, Kumar C, Sreedhar A. A split mouth randomized controlled study to evaluate the adjunctive effect of platelet-rich fibrin to coronally advanced flap in Miller's class-I and II recession defects. J Indian Soc Periodontol. 2013 Sep;17(5):631-6. doi: 10.4103/0972-124X.119281. PMID 24174758
- [Background] Nanditha S, Priya MS, Sabitha S, Arun KV, Avaneendra T. Clinical evaluation of the efficacy of a GTR membrane (HEALIGUIDE) and demineralised bone matrix (OSSEOGRAFT) as a space maintainer in the treatment of Miller's Class I gingival recession. J Indian Soc Periodontol. 2011 Apr;15(2):156-60. doi: 10.4103/0972-124X.84386. PMID 21976841